CLINICAL TRIAL: NCT01678352
Title: A Pilot Study to Evaluate the Effects of Imiquimod and Tumor Lysate Vaccine Immunotherapy for Adults With High Risk or Recurrent/Post-Chemotherapy WHO Grade II Gliomas
Brief Title: Imiquimod and Tumor Lysate Vaccine Immunotherapy in Adults With High Risk or Recurrent Grade II Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Frank Lieberman (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Frank Lieberman, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-136
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: High Risk WHO Grade II Glioma; Recurrent/Post-Chemotherapy WHO Grade II Glioma
Keywords: Glioma; Vaccine; Immunotherapy; WHO Grade II
MeSH Terms: conditions — Glioma; Lymphoma, Follicular | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients must have undergone surgery or biopsy alone (no postoperative radiation or chemotherapy) and have a baseline MRI scan (within 4 weeks of the first vaccine) that shows stable disease or regression (no progression from the initial surgery/biopsy).
  Interventions: Biological: Tumor Lysate Vaccine; Drug: Imiquimod
- Cohort 2 (Experimental): Patients received surgery or biopsy and radiation therapy (RT) (including fractionated external beam radiation therapy and/or stereotactic radiosurgery), which was completed ≥ 6 months prior to enrollment, and have a baseline MRI scan within 4 weeks prior to the first vaccine that shows stable disease or regression.
  Interventions: Biological: Tumor Lysate Vaccine; Drug: Imiquimod
- Cohort 3 (Experimental): Patients with recurrent WHO grade 2 glioma may have received prior external beam radiotherapy and/or chemotherapy. Patients with stable WHO grade 2 glioma must have had prior chemotherapy (at least one cycle of Temozolomide or PCV-based chemotherapy). With regard to the prior therapy in Cohort 3, patients may have had treatment for no more than 2 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy) or observation of stable disease. The intent therefore is that patients may have had 3 prior therapies (initial therapy and treatment for 2 relapses). If the patient had a surgical resection for relapsed disease, and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse.
  Interventions: Biological: Tumor Lysate Vaccine; Drug: Imiquimod

INTERVENTIONS:
Biological: Tumor Lysate Vaccine — Cohort 1 Cohort 2 Cohort 3
Drug: Imiquimod — Cohort 1 Cohort 2 Cohort 3
  Other Names: Aldara

SUMMARY:
This is a pilot study of a vaccination regime that is designed to efficiently induce anti-tumor T-cell responses in patients with WHO grade II glioma. The proposed regime with BTIC Lysate in combination with imiquimod, an FDA-approved immune response modifier will induce potent anti-glioma immune response with minimal or no toxicity.

DETAILED DESCRIPTION:
To determine the response rate and magnitude of CD8+ T-cell responses against the Imiquimod/BTIC lysate-based vaccines in post-vaccine PBMC using IFN- ELISPOT. ELISPOT assays indicate functional status of the antigen-specific T cells as cytokine-expression, and we are particularly interested in Type-1 (i.e. IFN expressing) T cell response. Therefore, IFN ELISPOT will be used as the primary assay for the immunological endpoint.

Using flow-cytometry, we will also evaluate the numbers of lymphocyte subsets such as CD4+ T cells, CD4+/Foxp3+ regulatory T cells in an exploratory manner. In addition, in participants who undergo surgical debulking of the progressing tumor, if the tumor tissue is available, infiltration of antigen-specific CTLs will be evaluated by flow cytometry of tumor-infiltrating lymphocytes with the Imiquimod/BTIC lysate-based vaccine-targeted GAA specific MHC-tetramers. In addition, serological responses will be evaluated with flow-cytometry of BTIC cells as well as western blotting. These plans (in this paragraph) are immunological evaluations; however, do not compose the primary endpoints due to their exploratory nature.

We will determine whether it is safe to administer Imiquimod/BTIC lysate-based vaccines in patients with grade II gliomas. Endpoints will therefore include incidence and severity of adverse events, using standard criteria as well as close clinical follow-up as would be performed normally in this group of participants following vaccinations. All reported or observed toxicities and adverse events at all clinic visits will be graded, documented and reported according to a standard toxicity table, the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 and 2: Age ≥18 year old with histologically diagnosed World Health Organization (WHO) grade II astrocytoma or oligoastrocytoma with "high-risk" factors - defined as:

  * age ≥ 40 with any extent resection;
  * age 18-39 with incomplete resection (post-op MRI showing >1cm residual disease, based on the maximum dimension of residual T2 or fluid-attenuated inversion-recovery [FLAIR] abnormality from the edge of the surgical cavity either laterally, anteroposteriorly, or superoinferiorly) or
  * age 18-39 with neurosurgeon-defined gross total resection (GTR) but the tumor size is ≥ 4 cm (the maximum preoperative tumor diameter, based on the axial and/or coronal T2 or FLAIR MR images) Cohort 3: Age ≥18 year old with histologically diagnosed WHO grade II glioma with recurrence
  * Karnofsky performance status ≥ 60%
  * Clinically stable and off corticosteroids for at least 4 weeks prior to study enrollment
  * Adequate organ function within 14 days of study registration including:
  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1.0 x 109/L, platelets ≥100 x 109/L; hemoglobin ≥ 8 g/dL
  * Hepatic: - Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age and SGPT (ALT) ≤ 2.5 x upper limit of normal (ULN) for age
  * Renal: Normal serum creatinine or creatinine clearance ≥60 ml/min/1.73 m2

Exclusion Criteria:

* History of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) that required systemic immunosuppression therapy and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immunosuppression)
* Any isolated laboratory abnormality suggestive of a serious autoimmune disease (e.g. hypothyroidism)
* Any conditions that could potentially alter immune function (AIDS, multiple sclerosis, diabetes, renal failure)
* Receiving ongoing treatment with immunosuppressive drugs, excluding those patients requiring dexamethasone for treatment of tumor-related edema
* Currently receiving any investigational agents or registration on another therapy based trial
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10; Primary Completion 2017-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Two Years
  The incidence and severity of adverse events associated with the vaccine regime will be assessed according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE), as follows:
  1. . Grade 3-5 vaccine related allergic reaction
  2. . Grade 3-5 organ toxicity (cardiac, dermatologic (excluding localized skin reaction), gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy and occurring within 28 days of vaccination and of any length in duration
  3. . Grade 2 -5 autoimmune reactions (such as hypothyroidism)
Induction of BTIC Lysate-specific T-cell response | Two Years
  We will determine the response rate and magnitude of immune response in post-vaccine peripheral blood mononuclear cells (PBMC) against the BTIC Lysate in response to this form of vaccine, using IFN-enzyme-linked immuno-spot (ELISPOT) assays.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lieberman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States